CLINICAL TRIAL: NCT06469047
Title: Relationship Between Serum N/OFQ and Acute Myeloid Cell Leukemia
Acronym: RBSNAAMCL
Status: Not yet recruiting | Type: Observational
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, professor, Second Hospital of Shanxi Medical University
Other Study IDs: Hanyi20240408
Record Dates: First submitted 2024-06-16; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: AML

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- the newly diagnosed group
  Interventions: Diagnostic Test: Enzyme-linked immunosorbent assay
- the relapsed group
  Interventions: Diagnostic Test: Enzyme-linked immunosorbent assay
- the complete remission group
  Interventions: Diagnostic Test: Enzyme-linked immunosorbent assay
- the control group
  Interventions: Diagnostic Test: Enzyme-linked immunosorbent assay

INTERVENTIONS:
Diagnostic Test: Enzyme-linked immunosorbent assay — Serum N/OFQ , IL-1β and NE levels were detected.

SUMMARY:
Patients diagnosed with acute myeloid leukemia in the Second Hospital of Shanxi Medical University were selected and divided into the newly diagnosed group, the relapsed group, the complete remission group as the experimental group, and the healthy physical examination subjects as the control group. The relationship between IL-1β, catecholamine and norkephalin in peripheral blood of the experimental group and the control group was observed. According to the literature, the experimental group was significantly higher than the control group. In the experimental group, the newly diagnosed group was higher than the relapse group, and the relapse group was higher than the complete remission group, and the correlation was positive, and the difference was statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* In accordance with adult acute myeloid leukemia (non-acute promyelocytic leukemia)The diagnostic criteria for AML in the Chinese Diagnosis and Treatment Guidelines (2017 edition); ②Leukocyte count ≤ 25×109/L;

  * No treatment has been received in the past 6 months.

    * None of the candidates are related and known this study, and sign the informed consent.

Exclusion Criteria:

* Patients who are allergic to the drugs used in this study;

  * People with mental illness or cognitive impairment;

    * Patients with infectious diseases; ④Patients with severe heart, liver, kidney and other organ function lesions; ⑤ Combined with other malignant swelling. The tumor.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the Second Hospital of Shanxi Medical University from June 2022 to November 2023
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
N/OFQ | 24 hours
  Serum N/OFQ levels
IL-1β | 24 hours
  Serum IL-1β levels
NE | 24 hours
  Serum NE levels

CONTACTS AND LOCATIONS:
Locations (1):
- Second Hospital of Shanxi Medical University, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No